CLINICAL TRIAL: NCT00148265
Title: Phase II/III Multicentre Randomised Clinical Trial of Laser Treatment Plus 4 mg Intravitreal Triamcinolone Injection to Reduce Diabetic Macular Oedema
Brief Title: A Multicentre Randomised Clinical Trial of Laser Treatment Plus Intravitreal Triamcinolone for Diabetic Macular Oedema
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Sydney (Other)
Collaborators: The University of Western Australia (Other); University of Melbourne (Other); Marsden Eye Specialists (Other)
Responsible Party: Professor Mark Gillies, Save Sight Institute, The University of Sudyney
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NHMRC project 352312
Record Dates: First submitted 2005-09-06; First posted 2005-09-07 (Estimated); Last update posted 2010-06-23 (Estimated); Status verified 2005-11

CONDITIONS: Diabetic Macular Oedema
Keywords: Diabetic macular oedema; Triamcinolone acetate; Intravitreal injection; Clinical trial; Laser treatment
MeSH Terms: interventions — Triamcinolone; Triamcinolone Acetonide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Triamcinolone acetate — Eyes assigned to IVTA received an intravitreal injection of 0.1 ml of Kenacort 40© [40mg/ml triamcinolone acetonide, Bristol-Myers Squibb pharmaceuticals, Australia] on the day of the baseline visual acuity measurement under sterile conditions in a minor procedures area as an outpatient procedure. Eyes assigned to placebo were prepared in the same way but had the barrel of the syringe without a needle pushed firmly against the eye to simulate an injection.
  Other Names: Kenacort 40©

SUMMARY:
This study is likely to identify an improved and economical treatment for diabetic macular oedema, one of the commonest causes of blindness both in Australia and the rest of the world.The specific aims of the study are to test the following hypotheses:

* That intravitreal triamcinolone followed by laser treatment results in a greater improvement in visual acuity than placebo followed by laser treatment of eyes with macular oedema secondary to diabetes;
* That intravitreal triamcinolone followed by laser treatment results in greater degree of resolution of macular oedema than placebo followed by laser treatment of eyes with macular oedema secondary to diabetes;
* That intravitreal triamcinolone followed by laser treatment results in a reduced requirement for further laser treatment to control diabetic macular oedema than placebo followed by laser treatment;
* That intravitreal triamcinolone followed laser has a manageable and acceptable safety profile in eyes with diabetic macular edema.

DETAILED DESCRIPTION:
A 25 fold increase in the risk of going blind on diagnosis of diabetes is one of the most daunting threats that people with diabetes face. Stimulated by several uncontrolled, anecdotal reports, we are already conducting a randomized clinical trial of intravitreal triamcinolone for the treatment of diabetic macular edema which is refractory to conventional laser treatment. The analysis of the 3 month data from this study has already unequivocally demonstrated that the treatment very significantly reduces or eliminates macular oedema in the short term and results in improved visual acuity. Thus intravitreal triamcinolone may represent the most significant development in the prevention of blindness in people with diabetes since the introduction of laser treatment. It is also a highly cost-effective intervention that can be administered by general ophthalmologists. The next question to be answered, which will be addressed directly by the present study, is whether there is a significant, synergistic beneficial effect when intravitreal steroids are combined with current therapy (laser).

This study represents the second major project to be undertaken by the Australian Retinal Collaboration (ARC). The ARC aims to set the highest attainable standards for investigator-initiated clinical research in retinal diseases in Australia. Having enrolled and treated more than the target of 120 patients, we are currently completing an RCT of laser induced chorioretinal anastomosis for central retinal vein occlusion, an innovative Australian concept for a severe and otherwise untreatable disease. The proposed study is likely to identify an improved and economical treatment for one of the commonest causes of blindness both in Australia and the rest of the world. Intravitreal triamcinolone is also an intervention which has generated intense interest internationally, and one for which members of the ARC are acknowledged pioneers.

Successful implementation of the study proposed, which is feasible, is highly likely to have an immediate and direct effect on the prevention of vision impairment and blindness in people with diabetes

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Diagnosis of diabetes mellitus types 1 or 2
* Diabetic macular oedema affecting the fovea in one or both eyes (phakic or pseudophakic) for which laser treatment is indicated in the opinion of the investigator
* Best corrected visual acuity of 19-68 letters (6/12 -6/120)
* Definite macular oedema on clinical examination involving the centre of the macula
* Retinal thickness > 250 micron in central 1mm subfield on OCT
* Investigator is comfortable deferring macular laser treatment for 6 weeks

Exclusion Criteria:

* Glaucoma which is uncontrolled or is controlled but with glaucomatous field defects
* Loss of vision due to other causes (e.g. age related macular degeneration, myopic macular degeneration, retinal vein occlusion)
* Macular oedema due to other causes including vitreous traction
* An ocular condition that would prevent visual acuity improvement despite resolution of oedema (such as foveal atrophy)
* Previous treatment IVTA within 6 months or with peribulbar TA within 3 months
* Cataract surgery within the last 6 months
* Retinal laser treatment within the last 4 months
* High risk PDR at baseline or laser therapy cannot be delayed for 6 weeks on retina
* History of herpes viral disease in study eye
* Media opacity including cataract that already precludes adequate macular photography and laser treatment, or cataract that is likely to preclude an adequate view within 2 years
* Known allergies to triamcinolone acetate
* Patient is already receiving systemic steroid treatment
* Intercurrent severe disease such as septicemia, any condition which would affect follow-up or photographic documentation (e.g. geographical, psycho-social)
* History of chronic renal failure requiring dialysis or renal transplant
* Blood pressure >180/110 mmHg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2005-04; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
The proportion of eyes showing an improvement of visual acuity by 10 letters on a LogMAR chart compared with the pre-injection level 24 months after treatment | 24 month
  At 24 months, improvement of ≥10 LogMAR letters was seen in 15/42 (36%) eyes treated with IVTA plus laser compared with 7/42 (17%) eyes treated with laser only (p=0.047, odds ratio 2.79, 95% CI, 1.01, 7.67).

SECONDARY OUTCOMES:
Number of laser treatments required for the treatment of macular oedema during the course of the study. | 24 month
  At least 1 retreatment was required in the second year of the study in 29/42 (69%) of IVTA plus laser treated eyes compared with 19/42 (45%) laser only eyes (p=0.187).
Change in retinal thickness demonstrated on optical coherence tomography (OCT) | 24 month
  There was no difference in the mean CMT (346.8μm ± 114.9SD vs 372.6μm ± 154.2SD, comparing IVTA plus laser vs laser only, p=0.349) or mean logMAR visual acuity (56.1 ± 15.7SD vs 54.5 ± 16.1SD letters, p=0.439).
The incidence of moderate or severe side effects related to the procedure of intravitreal injection or related to the drug | 24 month
  Cataracts were removed from 17/28 (61%) of phakic IVTA plus laser-treated eyes vs. 0/27 (0%) laser only eyes (p<0.001). Treatment for elevated intraocular pressure was required in 27/42 (64%) of the IVTA plus laser eyes compared with 10/42 (24%) laser only eyes (p<0.001)

CONTACTS AND LOCATIONS:
Overall Officials: Mark C Gillies, MBBS, PhD, Principal Investigator — Save Sight Institute, Deaprtment of Clinical Ophthalmology, University of Sydney; Ian L McAllister, MBBS, Principal Investigator — Lions Eye Institute, The University of Western Australia; Tien Wong, MBBS, PhD, Principal Investigator — Royal Victoria Eye & Ear Hospital, Department of Ophthalmology, University of Melbourne; Jennifer Arnold, MBBS, Principal Investigator — Marsden Eye Centre Parramatta
Locations (1):
- Save Sight Institute, Sydney/Sydney Eye Hospital Campus, University of Sydney, Sydney, New South Wales, Australia

REFERENCES:
- [Background] Sutter FK, Simpson JM, Gillies MC. Intravitreal triamcinolone for diabetic macular edema that persists after laser treatment: three-month efficacy and safety results of a prospective, randomized, double-masked, placebo-controlled clinical trial. Ophthalmology. 2004 Nov;111(11):2044-9. doi: 10.1016/j.ophtha.2004.05.025. PMID 15522370
- [Background] Larsson J, Zhu M, Sutter F, Gillies MC. Relation between reduction of foveal thickness and visual acuity in diabetic macular edema treated with intravitreal triamcinolone. Am J Ophthalmol. 2005 May;139(5):802-6. doi: 10.1016/j.ajo.2004.12.054. PMID 15860283
- [Result] Wickremasinghe SS, Rogers SL, Gillies MC, Zhu M, Wong TY. Retinal vascular caliber changes after intravitreal triamcinolone treatment for diabetic macular edema. Invest Ophthalmol Vis Sci. 2008 Nov;49(11):4707-11. doi: 10.1167/iovs.08-1678. Epub 2008 Jul 3. PMID 18599569
- [Result] Mohamed Q, Gillies MC, Wong TY. Management of diabetic retinopathy: a systematic review. JAMA. 2007 Aug 22;298(8):902-16. doi: 10.1001/jama.298.8.902. PMID 17712074
- [Result] Gillies MC, Islam FM, Zhu M, Larsson J, Wong TY. Efficacy and safety of multiple intravitreal triamcinolone injections for refractory diabetic macular oedema. Br J Ophthalmol. 2007 Oct;91(10):1323-6. doi: 10.1136/bjo.2006.113167. Epub 2007 Apr 3. PMID 17405800
- [Result] Gillies MC, McAllister IL, Zhu M, Wong W, Louis D, Arnold JJ, Wong TY. Pretreatment with intravitreal triamcinolone before laser for diabetic macular edema: 6-month results of a randomized, placebo-controlled trial. Invest Ophthalmol Vis Sci. 2010 May;51(5):2322-8. doi: 10.1167/iovs.09-4400. Epub 2009 Dec 17. PMID 20019369